CLINICAL TRIAL: NCT05421871
Title: Comparison of Spinal Stabilization Exercises Vs Maitland Mobilization Along With Laser Therapy in Non-Specific Low Back Ache
Brief Title: Comparison of Spinal Stabilization Exercises Vs Maitland Mobilization Along With Laser Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DPT/Batch-Fall17/509
Record Dates: First submitted 2022-05-05; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Low Back Ache
MeSH Terms: conditions — Low Back Pain | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spinal Stabilization Exercises (Experimental): Spinal Stabilization Exercises technique
  Interventions: Behavioral: Spinal Stabilization Exercises
- Maitland Mobilization Along With Laser Therapy (Experimental): Maitland Mobilization Along With Laser Therapy technique
  Interventions: Behavioral: Maitland Mobilization Along With Laser Therapy

INTERVENTIONS:
Behavioral: Spinal Stabilization Exercises — Spinal Stabilization Exercises technique
  Arms: Spinal Stabilization Exercises
Behavioral: Maitland Mobilization Along With Laser Therapy — Maitland Mobilization Along With Laser Therapy technique
  Arms: Maitland Mobilization Along With Laser Therapy

SUMMARY:
Comparison of Spinal Stabilization Exercises Vs Maitland Mobilization Along with Laser Therapy in Non-Specific Low Back Ache

DETAILED DESCRIPTION:
Comparison of Spinal Stabilization Exercises Vs Maitland Mobilization Along with Laser Therapy for finding the better method for the treatment of Non-Specific Low Back Ache

ELIGIBILITY:
Inclusion Criteria:

* Both male and female within the age range of 18-60 years.
* Visual analogue scale that scores 3 and higher.
* Non radiating low back pain

Exclusion Criteria:

* Patients with a history of spinal diseases and injury
* Spinal stenosis
* Degenerative changes
* Neuropathy
* Intervertebral disc collapse.
* Spinal discectomy
* Spinal laminectomy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Spinal Stabilization Exercises in Non-Specific Low Back Ache | 6 Months
  26 participants with the exercises include double knee to chest, single knee to chest, pelvic tilting,bridging and hamstring muscle stretching.(2) The stabilization exercises will be performed for 25 minutes. The patients will be educated on correct posture and starting positions for their exercises. Roland-Morris disability questionnaire to check the ovelall condition.

SECONDARY OUTCOMES:
Maitland Mobilization Along with Laser Therapy in Non-Specific Low Back Ache | 6 Months
  26 participants with the most commonly used Maitland technique is central posterior-anterior mobilization in which the therapist will perform 4 sets of mobilization for 30 seconds in grade I which will be administered to the three spinous processes around the most painful areas which will be followed by grade II with a rest interval of 30 seconds. Roland-Morris disability questionnaire to check the ovelall condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Zahra Medical complex Johar town, Laser spine center Model town, Laser spine center Johar town., Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No